CLINICAL TRIAL: NCT06932796
Title: Reducing Intersectional and HIV Stigma Among High Risk Women Who Use Drugs in Kazakhstan, Central Asia: A Multilevel Stigma Resistance and Enacted Stigma Reduction Intervention for Women and Providers
Brief Title: Project Orleu: Reducing Intersectional and HIV Stigma Among Health Care Providers and High Risk Women Who Use Drugs in Kazakhstan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Fogarty International Center of the National Institute of Health (NIH); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Brooke West, Associate Professor, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAU3129; R01TW012405 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Stigma, Social
Keywords: Intersectional Stigma; HIV; Linkage to Prevention and Care; Service Delivery; Women; Drug Use; Sex Work
MeSH Terms: conditions — Social Stigma; Sex Work

STUDY DESIGN:
Intervention Model Description: Pre/Post Design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Provider Training and Clinic Messaging (Experimental): Providers receive a 5-session stigma-free clinic training and anti-stigma messaging campaign materials to display in clinic.
  Interventions: Behavioral: Health Care Provider Stigma Training and Clinic-Based Messaging Campaign

INTERVENTIONS:
Behavioral: Health Care Provider Stigma Training and Clinic-Based Messaging Campaign — Providers in 10 HIV clinics participated in a 5 session anti-stigma health facility training focused on: 1) raising awareness about stigma and discrimination at the facility; and 2) changing attitudes and behaviors towards women who use drugs and/or trade sex; and 3) building a stigma-free clinic. Each of these clinics also received anti-stigma messaging materials (i.e., pamphlets, posters) to display in their clinics over a 6 month period. Providers received text-based message twice a month during this time to reinforce skills learned during trainings and to empower providers to be stigma change agents. Providers completed pre/post survey assessments.

SUMMARY:
Suboptimal linkage to and retention in HIV prevention and care is prevalent among high-risk women who use or inject drugs in both the US and globally, including high HIV incidence contexts like Kazakhstan; addressing HIV and intersectional stigma, especially from health care providers (HCP) within clinics, is necessary to increase engagement in the HIV care and prevention continuum. To address this challenge and increase HIV prevention and care, the proposed study will involve the design and assessment of the acceptability, feasibility, and usability of a three component, multi-level participatory intervention to promote stigma resistance/coping and reduce anticipated/internalized stigma among high-risk women who use drugs as well as to reduce enacted stigma among HCP in Kazakhstan, Central Asia. Results of this study will generate information in order to power a future preliminary effectiveness trial and will be unique in utilizing multilevel anti-stigma approaches for both high risk women who use drugs and HCP, all of which will have important implications for advancing HIV prevention and care engagement among highly stigmatized populations in diverse settings.

DETAILED DESCRIPTION:
Suboptimal linkage to and retention in HIV prevention and care is prevalent among high-risk women who use or inject drugs in both the US and globally, stemming, in part, from high levels of stigma. In Kazakhstan, increasing engagement in the HIV care and prevention continuum is a major public health goal, as the number of new HIV infections doubled from 2010 to 2017 and AIDS-related deaths increased by 32%. Among high-risk women who use drugs in this context, research has found that ~30% are HIV-infected and that they are less likely to test and receive care. Numerous studies have documented that experienced, anticipated and internalized stigma, especially from health care providers (HCP), are key barriers to HIV testing and treatment in global contexts. For high-risk women who use drugs, HIV and associated stigmas, specifically stigma related to sex and drug use, as well as gender discrimination, work independently and synergistically to inhibit access to HIV prevention and treatment; yet, there are no existing anti-stigma interventions designed and tested in Kazakhstan for this key population of women and that focus on HCP as sources of stigma. This study proposes to design and assess acceptability, feasibility, and generate information in order to power a preliminary effectiveness trial of a three component, multi-level participatory intervention to reduce HIV-associated and intersectional stigma - and thus increase access to HIV prevention and care. The first component is aimed at high-risk women and designed to increase stigma resistance/coping and reduce anticipated/internalized stigma via: a) crowdsourcing of anti-stigma messaging for HCP; and b) adaptation of an HCP training for optimal sexual health and healthcare engagement among high-risk women who used drugs. The second and third components, aimed at the HCP and other clinic staff and emerging from the execution of the first component, include: a) the resultant messaging campaign; and b) the training that will be delivered to HCP. Both the messaging campaign and the training components will be designed to reduce enacted stigma by HCP/staff (and thus experienced stigma among women) and increase stigma resistance and resilience among high-risk women who use drugs. All components will work synergistically to reduce enacted, experienced and internalized, intersectional stigma. The approach relies on evidence-based methods, including media campaigns, to reduce HCP enacted stigma, and integrates innovative methods, like crowdsourcing and participatory research, to increase stigma resistance. Results of this study will be unique in utilizing multilevel anti-stigma approaches for both high-risk women who use drugs and HCP and have important implications for advancing HIV prevention and care engagement among highly stigmatized populations globally and in the US.

ELIGIBILITY:
Inclusion Criteria:

* Providers (e.g., physicians, nurses, clinic directors, epidemiologists, outreach workers)
* Aged 18 years or older
* Currently employed part or full-time at an AIDS Center friendly clinic (city clinics focused on the provision of HIV and sexual health care).

Exclusion Criteria:

- Providers who are less than 18 years of age and/or do not work at an AIDS center friendly clinic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2024-08-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Provider HIV Enacted Stigma Measure | 6 months
  This 4-item measure is adapted from the "Measuring HIV Stigma and Discrimination among Health Facility Staff" questionnaire enacted stigma sub-scale. Across the 4 items, Likert-responses range from 1 (never observed) to 4 (always observed).

SECONDARY OUTCOMES:
Total Number of PrEP Prescriptions Issued to Clients | 6 months
  Through review of clinic-level administrative data, this study will measure the total number of prescriptions for PrEP over a 6-month period.
Total Number of Clients | 6 Months
  Through review of clinic-level administrative data, this study will measure the total number of clients over a 6-month period.

CONTACTS AND LOCATIONS:
Locations (1):
- Global Health Research Center for Central Asia, Almaty, Kazakhstan

IPD SHARING:
Plan to Share IPD: No
After further testing, we will share study protocols.